CLINICAL TRIAL: NCT04243512
Title: Time-restricted Eating in Cancer Survivorship: A Single-arm Feasibility Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Amber Kleckner, Research Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMLT19187
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-06

CONDITIONS: Cancer Survivorship

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time-restricted eating (Experimental): Participants will be asked to follow a TRE meal pattern for 14 consecutive days. Participants will be encouraged to consume food and beverages only within a 10-h time window for the 14-day intervention, with the exception of water, which will be encouraged at any time.
  Interventions: Behavioral: Time-restricted eating

INTERVENTIONS:
Behavioral: Time-restricted eating — Restrict food and beverage intake (except water) to a 10-hour window

SUMMARY:
The investigators will assess the feasibility of delivering a time-restricted eating (TRE) intervention among cancer survivors with fatigue.

DETAILED DESCRIPTION:
In this study, the feasibility of delivering a time-restricted eating (TRE) intervention among fatigued cancer survivors will be assessed. The participants will be asked to eat ad libitum only within a self-selected 10-h window each day for 14 days. The primary aim is to assess the adherence of the participants to the 10-h TRE intervention.

ELIGIBILITY:
Inclusion Criteria (Participants must...)

* Have completed adjuvant chemotherapy, surgery, and/or radiation for cancer at least 4 months and not more than 5 years prior to enrolling,
* Have a baseline level of fatigue, as determined by reporting a score of 3 or higher for the question, "In the last week, how bad was your worst fatigue on a scale from 0-10?"
* Be able to speak English,
* Be at least 18 years old,
* Be willing and able to adhere to study procedures, and
* Be able to provide written informed consent.

Exclusion Criteria (Participants must not...):

* Already eat all their food within a window that is 10 h or shorter most (6/7) days of the week,
* Be underweight, as defined as a body mass index ≤20.0 kg/m2.
* Not have surgery planned in the next month,
* Not have any contraindications to the proposed nutrition intervention as identified by
* their medical provider, their designee, or the study team (e.g., type 1 diabetes, risk for hypoglycemia, medication requirements, pregnancy, breastfeeding, recent history of an eating disorder),
* Not be taking insulin, or
* Be on enteral or parenteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmot Cancer Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kleckner AS, Altman BJ, Reschke JE, Kleckner IR, Culakova E, Dunne RF, Mustian KM, Peppone LJ. Time-restricted Eating to Address Cancer-related Fatigue among Cancer Survivors: A Single-arm Pilot Study. J Integr Oncol. 2022;11(5):379. Epub 2022 May 30. PMID 36131848

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Time-restricted Eating
Started | 39
Completed | 36
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Time-restricted Eating
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent of Days That Participants Adhere to the TRE Dietary Pattern
Description: Adherence will be assessed as the percent of days that each participant adheres to the 10-h TRE dietary pattern
Time Frame: 14 days
Measure: Mean (Full Range); unit: percent of days
Arm/Group | Time-restricted Eating
Number analyzed (Participants) | 36
percent of days | 90.1 [43 to 100]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Time-restricted Eating
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 2/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Time-restricted Eating (N=39)
headache (General disorders) | 1 (1)
insomnia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT04243512/Prot_SAP_000.pdf